CLINICAL TRIAL: NCT00842881
Title: Clinical Efficacy and Safety of Healing Stone Navel Belt in Patients With Primary Dysmenorrhea
Brief Title: A Trial for Evaluation of Clinical Efficacy and Safety of Healing Stone Navel Belt in Patients With Primary Dysmenorrhea
Acronym: Healingstone
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Healingstone Co., Ltd. (Industry)
Responsible Party: Mijin Park / Manager, Healingstone Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-01-001
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Primary Dysmenorrhea
Keywords: Healingstone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- a (No Intervention): healingstone
  Interventions: Device: Healingstone navel belt
- b (No Intervention): stone powder
  Interventions: Device: Healingstone navel belt

INTERVENTIONS:
Device: Healingstone navel belt — 6~8hours/day for 3months
  Other Names: Serial Number : HS-402

SUMMARY:
The purpose of this study is to determine whether Healing stone navel belt is safe and effective in the treatment of Primary Dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Age : female adults aged 15~45 years
* Subjects should diagnosed as primary dysmenorrhea, should have a primary dysmenorrhea at least a 1-day during menstrual.
* Subjects should have 21~42 days menstrual cycle.
* menstrual pain : primary dysmenorrhea at least a 1-day during menstruation is over 5 VAS(Visual Analogue Scale) without drug.
* Subjects must have no Serious internal medicine.
* Subjects must provide signed informed consent prior to participation in any study-related procedures

Exclusion Criteria:

* Subject that oral contraceptive taken within 3 months
* Pregnancy or lactation.
* Subject have contraceptive that secrete hormone.
* Secondary dysmenorrhea
* pelvis inflammatory disease patient
* Other diseases or characteristics judged by the investigator to be incompatible with the assessments needed in this study or with reliable instillation of the study.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 102 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-03 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
10cm VAS of pain(Dysmenorrhea) | 5months

SECONDARY OUTCOMES:
quality of life (SF-36) | 7months

CONTACTS AND LOCATIONS:
Overall Officials: EungGi Min, MD, Principal Investigator — DongGuk University Hosipital